CLINICAL TRIAL: NCT06445829
Title: Magnesium Sulfate Combined With Intraarticular Cocktail Injection for Analgesia After Simultaneous Bilateral Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202400399A3
Record Dates: First submitted 2024-06-02; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis, Knee
Keywords: intraarticular injection
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cocktail injection with Magnesium Sulfate (Experimental): Cocktail injection with Marcaine, Dexamethasone, normal saline and Magnesium Sulfate
  Interventions: Drug: Magnesium sulfate
- Cocktail injection without Magnesium Sulfate (No Intervention): Cocktail injection with Marcaine, Dexamethasone, and normal saline

INTERVENTIONS:
Drug: Magnesium sulfate — adding 300mg magnesium sulfate into cocktail injection
  Arms: Cocktail injection with Magnesium Sulfate

SUMMARY:
Total knee arthroplasty is a safe procedure with excellent outcome. In recent years, simultaneous bilateral total knee arthroplasty has become more popular. In views of enhanced recovery after surgery, intraarticular cocktail injection for pain control has been developed. However, the safety accumulation dose for simultaneous bilateral knee injection is still an issue. Recently, adding magnesium sulfate to intraarticular cocktail injection in unilateral total knee arthroplasty has been proved effective for prolong pain control. We tempt to conduct a double blinded study to evaluate that whether adding magnesium sulfate intraarticular cocktail injection to one of the knees in simultaneous bilateral total knee arthroplasty patient could effectively decrease pain score with less analgesia dose or not.

ELIGIBILITY:
Inclusion Criteria:

* bilateral knee advanced osteoarthritis or osteonecrosis who tend to receive simultaneous bilateral total knee arthroplasty

Exclusion Criteria:

* hypersensitivity to magnesium sulfate
* hypermagnesemia
* severe cardiac, hepatic or renal compromised

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
VAS score | day 0, day 1, day 2, day 3, day 7
muscle power | day 0, day 1, day 2, day 3
Straight leg raised test | day 0, day 1, day 2, day 3
active range of motion | day 0, day 1, day 2, day 3

SECONDARY OUTCOMES:
Magnesium level in blood | day 0, day 1
Calcium level in blood | day 0, day 1

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhao C, Wang L, Chen L, Wang Q, Kang P. Effects of magnesium sulfate on periarticular infiltration analgesia in total knee arthroplasty: a prospective, double-blind, randomized controlled trial. J Orthop Surg Res. 2023 Apr 14;18(1):301. doi: 10.1186/s13018-023-03790-w. PMID 37060089
- [Result] Wang Q, Zhao C, Hu J, Ma T, Yang J, Kang P. Efficacy of a Modified Cocktail for Periarticular Local Infiltration Analgesia in Total Knee Arthroplasty: A Prospective, Double-Blinded, Randomized Controlled Trial. J Bone Joint Surg Am. 2023 Mar 1;105(5):354-362. doi: 10.2106/JBJS.22.00614. Epub 2023 Mar 1. PMID 36856693